CLINICAL TRIAL: NCT04194931
Title: Study Evaluating the Safety and Efficacy With Sequential Infusion of Humanized CAR-T Cells of Anti-BCAM and Anti-CD19 Against Relapsed and Refractory Multiple Myeloma
Brief Title: Humanized CAR-T Cells of Anti-BCAM and Anti-CD19 Against Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, LiFei,M.D., Ph.D., M.D.,Ph.D., The First Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018028
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Relapsed and refractory multiple myeloma; CAR-T
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mixed BCMA/CD19 CAR-T Transfer (Experimental): Subjects with BCMA/CD19+ multiple myeloma will be infused with CD19-targeting CAR T Cells and BCMA-targeting CAR T Cells in one time or in parts
  Interventions: Biological: Autologous BCMA CAR-T cells and CD19 CAR-T cells

INTERVENTIONS:
Biological: Autologous BCMA CAR-T cells and CD19 CAR-T cells — Autologous BCMA CAR-T cells and CD19 CAR-T cells with average 1-5*10^6 cells/kg body weight,separately.

SUMMARY:
This is a single arm, open-label, single center study to evaluate the safety and efficacy of BCMA/CD19 CAR-T cells in patients with BCMA+，CD19+ relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
CD19 has been extensively evaluated as a therapeutic target for relapsed or refractory multiple myeloma by chimeric antigen receptor T cell therapy,this is a single arm, open-label, single center study to preliminary explore the safety, tolerability and cellular pharmacokinetics of Anti-BCMA and Anti-CD19 CAR-T cells in the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-70 years old
2. Estimated Survival time > 12 weeks
3. Relapsed and refractory multiple myeloma were confirmed by physical examination, pathological examination, laboratory examination and imaging
4. Chemotherapy failure or recurrent multiple myeloma
5. Glutamic-pyruvic transaminase, glutamic oxalacetic transaminase< 3 fold of normal level
6. Bilirubin<2.0mg/dl
7. Karnofsky Performance Status>50% at the time of screening
8. Adequate pulmonary, renal, hepatic, and cardiac function
9. Fail in autologous haemopoietic stem cell transplantation
10. Not suitable for stem cell transplantation conditions or abandoned due to conditions
11. Free of leukocytes removal contraindications
12. Voluntarily join CAR-T clinical trial ,Understand and sign written informed consent

Exclusion Criteria:

1. The patient is a pregnant or breastfeeding woman, or is a woman with a pregnancy plan within six months
2. Patients have infectious diseases (such as HIV, active tuberculosis, etc.)
3. The patient is an active hepatitis B or hepatitis C infection
4. Feasibility assessment proves that the efficiency of transduction of lymphocyte is below 10% or the lymphocyte cannot be propagated
5. Abnormal vital signs
6. Subjects with mental or psychological illness who cannot be combined with treatment and efficacy evaluation.
7. Highly allergic constitution or history of severe allergies, especially allergy to interleukin-2
8. General infection or local severe infection, or other infection that is not controlled
9. Dysfunction in lung, heart, kidney and brain
10. Severe autoimmune diseases
11. Other symptoms that are not applicable for CAR-T

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 2 year
  Assessment of ORR (ORR = sCR+CR+VGPR+PR ) at 1 months of treatment
minimal residual disease（MRD） | 2 year
  Assessment of MRD negative overall response rate at 3 months of treatment
Progression-free survival (PFS) | 2 year
  Assessment of Progression-free survival (PFS) at 6 months of treatment
Overall survival (OS) | 2 year
  Assessment of overall survival (OS) at 6 months of treatment

SECONDARY OUTCOMES:
Safety (incidence of adverse events defined as dose-limited toxicity) | Study treatment until Week 24
  Occurrence of study related adverse events defined as NCI CTCAE 4.0 > grade 3 possibly, probably, or definitely related to study treatment.
Expression of CD19 CART cells | 2 year
  Expression of CD19 CART cells in blood, bone marrow by Quantitative Polymerase Chain Reaction (q-PCR) and by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nangchang University, Nanchang, Jiangxi, China